CLINICAL TRIAL: NCT04130685
Title: Donor-Derived Cell-Free DNA for Surveillance in Simultaneous Pancreas and Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: 19073007
Record Dates: First submitted 2019-10-07; First posted 2019-10-17 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Pancreas Transplant Rejection; Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Allosure Test — Venous Blood Draw

SUMMARY:
The AlloSure test is approved by the Centers for Medicare & Medicaid Services (CMS) for use in Medicare patients to assess the probability of allograft rejection in kidney transplant patients. The pivotal DART study discusses the use of the non-invasive AlloSure test to measure donor derived cell-free DNA (dd-cfDNA) and the Allosure test can by used to discriminate active rejection in renal transplant patients. Pancreas allograft rejection still remains a major clinical challenge and is a primary cause of death censored pancreas allograft loss. Pancreas transplant rejection is diagnosed by biopsy, however it is not commonly performed because of the complications such as pancreatic leak, graft loss and patient death. Currently at Rush surveillance biopsy of the pancreas are not performed routinely due to the above risks.

At RUMC, patients are followed post-transplant with series of labs at set intervals that include lipase, DSA, C-Peptide, and GAD65 for surveillance of rejection

The AlloSure test was introduced for routine use in kidney transplant recipients at Rush University Medical Center in October 2017, after CMS approval and then as part of the KOAR Study in May of 2018. AlloSure test has been included as part of the routine labs for surveillance of rejection in pancreas transplant recipients at RUMC since September 2018 after it was approved for compassionate use. The addition of AlloSure has helped to improve surveillance of rejection in pancreas transplant recipients and has reduced the need for the kidney biopsy as a surrogate marker of rejection in the pancreas.

Our goal is to determine if AlloSure can be used for surveillance for rejection in recipients of Simultaneous Pancreas and Kidney (SPK) Transplant recipients.

DETAILED DESCRIPTION:
This is a prospective and retrospective cohort study of recipients of simultaneous pancreas and kidney transplant recipients (SPK).

New SPK transplant recipients and previous SPK transplant recipients from September 2012 will be enrolled in the study, expected duration of participation will therefore range from a minimum of 1 year to a maximum of 5 years for each participant.

The visits are incorporated into the current standard of care in our program and no extra visits are required. Mobile draw for AlloSure can be obtained if the patient is not due for a visit when the AlloSure draw is due.

AlloSure labs will be drawn on all new SPK patients and results obtained as well as retrospective results that have already been received on past SPK recipients. The AlloSure will be added to the standard of care schedule for all SPK patients.

The schedule will be the following:

For newly transplanted patients, AlloSure will be checked at 14 days post-transplant

For all subjects:

From 1 month to 12 months post transplant: AlloSure will be obtained monthly with their transplant date as the reference time point

From 12 months to 36 months: AlloSure will be obtained every 3 months

From 36 months to 60 months: AlloSure will be obtained every 6 months.

AlloSure may be obtained more frequently than the above schedule, with other clinical data or allograft biopsy, if there is graft dysfunction or suspicion for rejection.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* New SPK transplant recipients
* SPK recipients from September 2012 with functioning kidney and pancreas, not on dialysis and/or insulin

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Unwilling to participate in research study
* Recipients of other solid organ transplants apart from the SPK
* Recipients of pancreas and kidney allografts from separate donors
* Recipients with SLE
* Patients who have received a bone marrow transplant
* Recipients of a transplant form a monozygotic twin
* Patients who are pregnant
* Patients below the age of 18 years
* SPK recipient on insulin at enrolment
* SPK recipient on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of Simultaneous Pancreas and Kidney (SPK) transplant since 2012 and above the age of 18 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To determine median AlloSure level in SPK recipients with stable allograft function | Median allosure level collected from two weeks post transplant up until 36 months post transplant.
  Percentage of dd-cfDNA (AlloSure) level in blood samples of recipients of kidney and pancreas transplant.

SECONDARY OUTCOMES:
The Allosure levels will be measured in the setting of rejection. | Throughout study completion, which is three years from date of transplant.
  Determine AlloSure levels at time of rejection
To determine the Allosure level post transplant | Throughout study completion, which is three years from date of transplant.
  AlloSure level

CONTACTS AND LOCATIONS:
Overall Officials: Oyedolamu Olaitan, MBBS, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cell-Free DNA and Active Rejection in Kidney Allografts. — https://pubmed.ncbi.nlm.nih.gov/28280140/